CLINICAL TRIAL: NCT04787679
Title: Image-guided Computational and Experimental Analyses of Fractured Patient's Bone (GAP)
Acronym: GAP
Status: Recruiting | Type: Observational
Sponsor: Laura Maria Vergani (Other)
Collaborators: Ospedale San Donato (Other)
Responsible Party: Sponsor-Investigator, Laura Maria Vergani, Professor, Politecnico di Milano
Organization: Politecnico di Milano (Other)
Other Study IDs: Polimi_Galeazzi_GAP
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis; Fragility Fracture
Keywords: lacunae; damage models; micro-cracks; synchrotron; numerical models
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Waste materials from human femoral heads collected after hip replacement surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoporotic patients: Osteoporotic patients, age > 18 years old
  Interventions: Procedure: Hip replacement surgery
- Non osteoporotic patients: Non osteoporotic patients, age > 18 years old
  Interventions: Procedure: Hip replacement surgery

INTERVENTIONS:
Procedure: Hip replacement surgery — After hip replacement surgery the sponsor obtains femoral head samples for the study

SUMMARY:
Due to the increase in the average age of the population, the projections on the number of age-dependent bone fractures appear to be constantly increasing.

They are mainly due to bone pathologies, including osteoporosis. The latter leads to a reduction in bone mineral density and deterioration of the micro-architecture, with a consequent increase in bone fragility. However, the mechanisms of damage at the micro-scale have not yet been elucidated and there is no universally recognized damage criterion. Recent research has evaluated the importance of implementing computational models to study the influence of bone gaps, canaliculi and microporosities on the propagation of damage. These models need to be validated through experimental tests, still lacking, in particular on human bones, in the current scientific landscape. Once the experimental validation of computational models has been developed, it will be possible to introduce new fracture indices at the micro-scale, useful for a preventive diagnosis of osteoporosis.

DETAILED DESCRIPTION:
The study of the mechanisms of bone damage, which occur at the multiscale, is of fundamental importance for the understanding of fracture processes. In particular, age-related fractures are continuously increasing due to the increase in average age and widespread diseases such as osteoporosis. They result in high economic burdens, morbidity (including psychological, e.g., frailty), and increased mortality. In order to reduce the impact of bone fractures on health and economy, early diagnosis is the key. In this context, one must consider that bone is characterized by a complex hierarchical structure. Both the cortical and trabecular sections consist of micrometric lamellae, composed of collagen fibrils, within which osteocytes are found. They reside in sub-micrometer cavities called lacunae, which are connected by a dense network of canaliculi. At the nanoscale, the fibrils consist primarily of collagen and hydroxyapatite crystals. This complex architecture is reflected in fracture patterns: damage, in fact, occurs at the multiscale. However, fracture patterns and their associated physical phenomena are still not understood, especially at the microscale.

Recently, microscale imaging techniques have been combined with subject-specific numerical models, which are able to calculate local values of bone stress and strain. Preliminary studies have focused on evaluating a possible interaction between micro-cracks and microstructural porosity. This particular research focuses on the lacunar network, which is presumed to significantly affect bone resistance to fracture although the actual role of the lacunar network is not yet elucidated. First, lacunae are areas of stress concentration, which apparently lead to weakening of the bone structure. However, in most cases, the lacunae make a positive contribution to toughness by deflecting the crack front. The connection between the lacunae, determined by the network of canaliculi, is also reduced in osteoporotic subjects, preventing the slowing of damage. In this sense, bone can be considered a damage tolerant material. Donaldson et al developed computational models and estimated a threshold for microdamage initiation and propagation. They used computerized micro-tomography of murine femurs and evaluated the influence of different algorithms on the propagation of in-silico damage. Further results showed that the damage always occurs on the surfaces of blood vessels or porosities and does not instead start from the lacunae. However, further simulations and models would be needed to verify the effectiveness of the damage models.

Computational damage models also require experimental validation. Preliminary studies have been conducted in two main directions: in-vivo imaging and image-guided failure assessment (IGFA) techniques. The first approach allows nondestructive monitoring of bone damage in living animals. The second approach, implemented by A. Levchuk et al. (8), shows enormous potential by allowing the study of microcrack initiation and propagation with sub-micrometer resolution, but only on small animals.

The current research for the first time wants to perform tests on human bone samples applying IGFA techniques.

Despite several studies on the characterization of damage models at the micro-scale, a validation of computational models of fracture on human subjects is still lacking. In addition, the role of morphological features at the micro-scale in samples is still unknown.

These micro-scale studies could improve clinical understanding of bone fracture and prediction of fracture risk. Currently, clinicians use bone mineral density, which is a macro-scale parameter, as the most common predictor of bone fracture. However, recent studies demonstrate the importance of a thorough characterization of the geometric and morphologic characteristics of the microarchitecture.

OBJECTIVES

General Objective The study aims at the experimental validation of computational models of bone damage at the micro-scale. The general objective is pursued by controlled damage in a micro-compression machine on human bone samples from femoral head. The machinery is placed inside a synchrotron.

Primary Objective The primary objective of the present study is to evaluate the difference in the attraction of bone damage with respect to gaps in the two groups considered (osteoporotic and non-osteoporotic) following micro-compression testing.

The discriminating parameter chosen turns out to be the number of bone gaps encountered by micro-damage. We expect to observe an effect size of 0.4 between the two groups with respect to the chosen parameter.

Secondary Objectives

* Determination of the role of gaps, canaliculi and other bone microstructures in damage. Human bone samples are scanned by micro-tomograph for the definition of microstructural morphological parameters and the realization and analysis of numerical models.
* Validation of these numerical models of damage by micro-compression tests carried out in situ in a synchrotron of adequate resolution
* Quantification of damage in human bone samples affected by osteoporosis
* Definition of micro-scale fracture indices, useful for the early diagnosis of osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Age: >=18 years
* primary hip replacement
* Signature of informed consent
* Patients who have a routine preoperative CT scan

Exclusion criteria:

* Patients unrelated to the inclusion criteria of this study
* Bone disease (non-osteoporotic) such as to invalidate sample analysis, including but not limited to genetic disorders and bone tumors
* Patients with contralateral hip replacement and/or other synthetic means in the contralateral hip
* Patients with synthesis devices in the hip of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of 52 subjects, 26 of whom are prosthetic and have osteoporosis detectable by preoperative computed tomography (CT) scan and 26 prosthetic whose CT scan does not indicate the presence of osteoporosis.
  The classification of the two groups will be made exclusively by analysis of routine preoperative CT scans according to standard radiological classification.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2028-08-09 (Estimated)

PRIMARY OUTCOMES:
Number of lacunae interested by damage | six months
  We expect to observe difference in osteoporotic and non osteoporotic samples interested or not by the damage

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Zagra, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Miano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided